CLINICAL TRIAL: NCT01338662
Title: A 10-year Observational Study of the Incidence of Dyskinesia in Patients With Early Parkinson's Disease Who Were Treated With Amantadine or Dopamine Agonist
Brief Title: Comparison of the Incidence of Dyskinesia in Parkinson's Disease Who Were Treated With Amantadine or Dopamine Agonist
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Other Study IDs: H-1009-057-332
Record Dates: First submitted 2011-04-05; First posted 2011-04-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A-1: * study enroll number 3n+1 (N=0,1,2...)
  * initial treatment- amantadine
  * add levodopa when the patient become to need further treatment.
- Group A-2: * study enroll number 3n+2 (N=0,1,2...)
  * initial treatment: amantadine
  * add dopamine agonist when the patient become to need further treatment.
- Group B: * study enroll number 3n+3 (N=0,1,2...)
  * initial treatment: dopamine agonist
  * add levodopa when the patient become to need further treatment. but cannot use amantadine

SUMMARY:
The purpose of this study is to compare the onset time and severity of dyskinesia in amantadine or Dopamine agonist initial treated groups in Parkinson's disease.

DETAILED DESCRIPTION:
1. Dopamine agonist can delay the risk of dyskinesia by initiating treatment rather than levodopa. Amantadine is typical antidyskinetic drug. There is no data about comparison of risk of dyskinesia in amantadine and dopamine agonist by initiating treatment.
2. Prospective , randomized, open label study compare the onset time and severity of dyskinesia between groups randomized assigned order of amantadine and dopamine agonist

ELIGIBILITY:
Inclusion Criteria:

* 30<age<60
* IPD
* H & Y<3

Exclusion Criteria:

* previous dopaminergic medication history
* dyskinesia
* Parkinson plus
* clinically significant or unstable medical or surgical condition

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: outpatient clinic in SNUH
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-05; Primary Completion 2020-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
dyskinesia onset | up to 10 years from the start of durg (Amantadine or dopaimine agonsit)
  observe duration of onset of dyskinesia from initial treatment observe until 10 years

SECONDARY OUTCOMES:
UPDRS, severity of dyskinesia between groups | observe duration of onset of dyskinesia from initial treatment
  observe duration of onset of dyskinesia from initial treatment observe until 10 years compare the UPDRS and severity of dyskinesia between groups

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Beom S Jeon, Seoul, South Korea

REFERENCES:
- [Background] Rascol O, Brooks DJ, Korczyn AD, De Deyn PP, Clarke CE, Lang AE. A five-year study of the incidence of dyskinesia in patients with early Parkinson's disease who were treated with ropinirole or levodopa. N Engl J Med. 2000 May 18;342(20):1484-91. doi: 10.1056/NEJM200005183422004. PMID 10816186
- [Background] Montastruc JL, Rascol O, Senard JM, Rascol A. A randomised controlled study comparing bromocriptine to which levodopa was later added, with levodopa alone in previously untreated patients with Parkinson's disease: a five year follow up. J Neurol Neurosurg Psychiatry. 1994 Sep;57(9):1034-8. doi: 10.1136/jnnp.57.9.1034. PMID 8089666